CLINICAL TRIAL: NCT03464643
Title: A Prospective Study Comparing the Outcomes of Single Embryo Culture Versus Group Culture in Preimplantation Genetic Testing Cycles
Brief Title: A Prospective Study Comparing the Outcomes of Single Versus Group Culture in Preimplantation Genetic Testing Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reproductive & Genetic Hospital of CITIC-Xiangya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KYXM-20180307
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Embryo Culture
MeSH Terms: interventions — Embryo Culture Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single embryo culture (Other): Embryo is cultured individually in 25 ul media
  Interventions: Other: embryo culture
- Group embryo culture (Other): 2-3 Embryos are group cultured in 50 ul media
  Interventions: Other: embryo culture

INTERVENTIONS:
Other: embryo culture — Single embryo culture means only one embryo is cultured in one drop, and the group culture refers to culture of 2-5 embryos in one drop. The main advantage of group culture may be secreting some paracrine cytokines by embryos and benefit each other; and the possible disadvantage of group culture is that embryo secreting of some harmful substances which accumulated to a certain extent will damage the developmental potential of embryos. The advantages and disadvantages of single embryo culture are contrary to group culture.

SUMMARY:
The aim of this study is to analyze whether there is difference in the effect of single embryo culture and group culture in preimplantation genetic screening (PGS) cycle, and provide reference for the feasibility of the clinical application of medium-based noninvasive PGD. This prospective study prepares for more than 1,000 normal fertilized zygotes in each group over one year period. For the recruited patients, all normal fertilized zygotes were randomly allocated into two groups: cultured individually in 25 ul media or 2-3 embryos cultured together in 50 ul media. The blastocyst formation rates, aneuploid rates, clinical pregnancy rates, implantation rates and miscarriage rates will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients treated by preimplantation genetic diagnostic / screening cycles

Exclusion Criteria:

* number of normal fertilization zygotes is less than 6

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 236 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2019-01-23 (Estimated); Study Completion 2019-09-23 (Estimated)

PRIMARY OUTCOMES:
high quality blastocyst formation rate | 6 days after fertilization
  number of blastocysts with high quality divided by number of zygotes with normal fertilization

SECONDARY OUTCOMES:
embryo euploid rate | about one month after blastocyst biopsy
  number of euploid blastocysts divided by all blastocysts detected
embryo implantation rate | about three to six months after blastocyst biopsy
  number of gestational sacs divided by number of embryo transferred

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojuan Wang, Doc, Principal Investigator — Reproductive and Genetic Hospital of Citic-xiangya
Locations (1):
- Reproductive and Genetic Hospital of Citic-xiangya, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided